CLINICAL TRIAL: NCT00139048
Title: A Randomised Controlled Trial of an On-line Decision Aid for Women Aged 40 Considering Whether to Have Screening Mammograms to Evaluate the Change in Knowledge Regarding Mammography Screening.
Brief Title: Australian Screening Mammography Decision Aid Trial: A Decision Aid for Women Aged 40 Thinking About Starting Mammography Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ASMDAT40
Record Dates: First submitted 2005-08-28; First posted 2005-08-30 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Knowledge of Mammography Screening
Keywords: informed choice; shared decision making; decision aid; mammography screening; decision support
MeSH Terms: interventions — Decision Support Techniques

INTERVENTIONS:
Behavioral: Decision Aid

SUMMARY:
Women who access the website, are aged between 38-45 years and are considering screening mammograms will be randomized to either the Decision Aid (a booklet providing information and exercises to help them to make a decision about whether to having screening mammograms) group or the Control Group. The Decision Aid group will first read the decision aid, and then will be asked some demographic and knowledge questions. The control group will be asked the demographic and knowledge questions only. The control group will have access to the Decision Aid after they have completed the questions

ELIGIBILITY:
Inclusion Criteria:

* female
* aged between 38-45
* have access to the internet

Exclusion Criteria:

-

Ages: 38 Years to 45 Years | Sex: Female
Age Groups: Adult
Enrollment: 200
Dates: Start 2005-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Assess the change in knowledge about the issues involved in screening mammography in women who have read the decision aid.

SECONDARY OUTCOMES:
elicit womens views on the decision aid including ease of use, content and presentation of information,
assess the differences in intention to screen
assess the impact of the decision aid on informed choice

CONTACTS AND LOCATIONS:
Overall Officials: Alex Barratt, Principal Investigator — Screening and Test evaluation programme, School of Public Health, University of Sydney
Locations (1):
- University of Sydney, Camperdown, New South Wales, Australia